CLINICAL TRIAL: NCT05575167
Title: The Effectiveness of Single or Repeat Zoledronate Infusion Versus Oral Alendronate in Consolidating the Bone Accrual Achieved With Denosumab: a Study Organised by the European Calcified Tissue Society
Brief Title: Single or Repeat Zoledronate Versus Alendronate Following Denosumab (EUROpean Denosumab Effects Consolidation Study)
Acronym: EURODEC
Status: Recruiting | Type: Observational
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Consultant of endocrinology; in charge of the Department of Metabolic Bone Diseases, 424 General Military Hospital
Other Study IDs: EURODEC
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Zoledronic Acid; Alendronate; Calcium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples for bone markers measurements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- single Zol group: postmenopausal women treated with denosumab for 3 or more years who will reach osteopenia with denosumab and will receive a single zoledronate infusion (5mg) at 6 months after the last denosumab dose
  Interventions: Drug: Zoledronate or Alendronate
- double Zol group: postmenopausal women treated with denosumab for 3 or more years who will reach osteopenia with denosumab and will receive two zoledronate infusions (5mg) at 6 and 12 months after the last denosumab dose
  Interventions: Drug: Zoledronate or Alendronate
- ALN group: postmenopausal women treated with denosumab for 3 or more years who will reach osteopenia with denosumab and will receive alendronate 70mg orally weekly for 12 months
  Interventions: Drug: Zoledronate or Alendronate

INTERVENTIONS:
Drug: Zoledronate or Alendronate — infusion (for zoledronate) or oral digestion (for alendronate)
  Other Names: Calcium and vitamin D supplementation

SUMMARY:
A 24-month prospective, open-label, randomized, multicenter, multinational, non-inferiority pragmatic clinical trial evaluating zoledronate single or double infusion versus oral alendronate following denosumab

DETAILED DESCRIPTION:
125 postmenopausal women treated with Dmab for 3 or more years who will reach osteopenia with denosumab will be randomized into three groups: i) zoledronate infusion (5mg) at 6 months after last Dmab dose (single Zol group) ii) zoledronate infusion (5mg) at 6 and 12 months after last Dmab dose (double Zol group) iii) alendronate 70mg orally weekly for 12 months (ALN group) All women will receive no further treatment during the 2nd year of the study.

Participating centers: ECTS affiliated bone centers

Endpoints: Primary: BMD changes at the lumbar spine at 12 months. Secondary: i) BMD changes at the lumbar spine at 24 months; ii) BMD changes at the non-dominant femoral neck and total hip at 12 and 24 months; iii) changes at levels of bone turnover markers throughout the study; iv) incident fractures: vertebral (clinical and morphometric identified on VFA scans) and non-vertebral; v) clinical parameters: height change, VAS for back pain, and use of analgesics

ELIGIBILITY:
Inclusion Criteria:

• Postmenopausal women treated with denosumab for 3 or more years who will reach osteopenia

Exclusion Criteria:

* a bone disease other than postmenopausal osteoporosis
* use of medications other than bisphosphonates or SERMS affecting bone metabolism during the last 12 months before entering the study
* creatinine clearance <60 mL/min/1.73 m2
* liver failure
* any type of cancer
* uncontrolled endocrine diseases
* serum 25-hydroxy vitamin D (25-OHD) concentrations lower than 20 ng/mL (50 nmol/L)

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Study Population: Postmenopausal women treated with denosumab
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
lumbar spine BMD | 24 months
  BMD changes at the lumbar spine at 12 and 24 months

SECONDARY OUTCOMES:
femoral neck BMD | 24 months
  BMD changes at the non-dominant femoral neck and total hip at 12 and 24 months
P1NP | baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  bone turnover (formation) marker
CTx | 24 months
  bone turnover (resorption) marker
fracture | 24 months
  incident fractures: vertebral (clinical and morphometric identified on VFA scans) and non-vertebral
height | 24 months
  loss of height

CONTACTS AND LOCATIONS:
Overall Officials: Willem Lems, Prof, Principal Investigator — ECTS Clinical Action Group
Locations (9):
- Univ. Lille, CHU Lille, Lille, France
- Greece (4):
  - 251 Hellenic Airforce and VA General Hospital, Athens
  - First Department of Propaedeutic and Internal Medicine, Medical School, National and Kapodistrian University of Athens, Athens
  - , KAT General Hospital, Athens
  - 424 General Military Hospital, Thessaloniki
- Italy (4):
  - Fondazione IRCCS Cà Granda-Ospedale Maggiore Policlinico, Milan
  - Campus Bio-Medico University, Roma
  - Department of Medicine, Surgery and Neurosciences, University of Siena, Siena
  - University-Hospital S. Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: Undecided